CLINICAL TRIAL: NCT07355114
Title: Robotic-assisted Unilateral Nephrectomy for Autosomal Dominant Polycystic Kidney
Brief Title: Robotic vs Open Nephrectomy for ADPKD
Acronym: ADPKDR-O
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Matteo Ravaioli, Professor, Director of Unit ''Chirurgia addominale nell'insufficienza d'organo terminale e nei pazienti con trapianto d'organo'', University of Bologna
Other Study IDs: ADPKDR-O
Record Dates: First submitted 2025-12-16; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Open nephrectomy: Unilateral Nephrectomy for ADPKD
- Robotic Nephrectomy: Unilateral Robotic nephrectomy for ADPKD with Hugo RAS System

SUMMARY:
The goal of this observational prospective cohort study is to evaluate the feasibility, safety, and postoperative outcomes of robotic-assisted unilateral native nephrectomy using the Medtronic Hugo™ RAS system compared with the open surgical approach in patients with autosomal dominant polycystic kidney disease (ADPKD)

The main question(s) it aims to answer are:

Is robotic-assisted unilateral nephrectomy with the Hugo™ RAS system feasible and safe in patients with ADPKD? Does robotic-assisted nephrectomy provide comparable or improved postoperative outcomes (e.g., complications, transfusion rates, length of hospital stay) compared with open nephrectomy? Researchers will compare robotic-assisted unilateral nephrectomy (Hugo™ RAS) with open unilateral nephrectomy to see if the robotic approach results in similar morbidity with shorter hospital stay, despite longer operative times.

Participants are adult patients with ADPKD undergoing unilateral native nephrectomy at a single tertiary transplant center, most of whom have end-stage renal disease and are candidates for or recipients of kidney transplantation. Both male and female patients were included; patients undergoing bilateral nephrectomy were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients who underwent unilateral nephrectomy for ADPKD

Exclusion Criteria:

* Patients who underwent bilateral nephrectomy for ADPKD were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients who underwent unilateral nephrectomy for ADPKD (Robotic with HUGO RAS System or open)
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Mortality by 90 day | By 90 days
  Mortality by 90 day

SECONDARY OUTCOMES:
Postoperative complications | By 90 days
  Postoperative complications described by Clavien-Dindo Classification

OTHER OUTCOMES:
Feasibility and safety of robotic-assisted native radical nephrectomy with Hugo RAS ™ in patients with ADPKD | Preoperative outcome measure: recorded at baseline Perioperative outcomes measure: perioperative/periprocedural Postoperative outcomes: up to 90 days after surgery. Follow up: through study completion
  Data were collected prospectively and retrospectively analyzed. Preoperative variables included demographics, presence of ERSD, history of previous abdominal surgery or previous transplant (liver, kidney or other), preoperative dialysis and type of dialysis (peritoneal or hemodialysis), comorbidities, Charlson Comorbidity index (Charlson-CI), American Society of Anesthesiologists (ASA) score, preoperative creatinine, hemoglobin, hematocrit and eGFR (calculated following the CKD-EPI equation [12]), kidney dimension measured on preoperative CT scan (cranio-caudal, antero- lateral and lateral length) and kidney volume. Perioperative and postoperative variables included operative time, the need of intraoperative and postoperative blood transfusion, intraoperative complications, drop in hemoglobin , the need of postoperative dialysis, complications (defined as major if Clavien-Dindo grade >2 )
Haemoglobin drop | Day 1
  Haemoglobin difference betweeen Baseling Haemoglobin in g/dl a and I POD hb
Operative time | Perioperative/Periprocedural
  Time in minutes from incision to skin closure

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: No